CLINICAL TRIAL: NCT01151865
Title: A Randomised, Double-blind, Multi-centre Placebo Controlled Trial of Dexmedetomidine for Patients With Agitation and Delirium in the Intensive Care Unit
Brief Title: Dexmedetomidine to Lessen Intensive Care Unit (ICU) Agitation
Acronym: DahLIA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Austin Health (Other Government)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, GLENN EASTWOOD, Associate Professor, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H2010/03891
Record Dates: First submitted 2010-06-18; First posted 2010-06-29 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Delirium
Keywords: Delirium; Intensive Care Unit; Dexmedetomidine
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine will be administered intravenously as a maintenance infusion of 0.2 to 1.5 mcg/kg/hour, commencing at 0.5 mcg/kg/hour and titrated according to effect, for as long as deemed necessary by the treating physician. Specifically, the study medication may be (as recommended by the manufacturer) continued after extubation, and if discontinued may be restarted at any time up until ICU discharge. The clinician will have the option of using a loading dose of 1.0 mcg/kg IV over 20 minutes, as recommended by the manufacturer.
  Bedside nursing staff will adjust drug infusion rates as necessary, in consultation with the treating physician, aiming to achieve a Riker Sedation-Agitation Scale 20 score of 4.
  Interventions: Drug: Dexmedetomidine
- Saline placebo (Placebo Comparator): An identical syringe to that in the intervention arm, but which does not contain dexmedetomidine, will be provided. The initial rate of infusion and subsequent adjustments will be the same as in the dexmedetomidine group.
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be administered intravenously as a maintenance infusion of 0.2 to 1.5 mcg/kg/hour, commencing at 0.5 mcg/kg/hour and titrated according to effect, for as long as deemed necessary by the treating physician. Specifically, the study medication may be (as recommended by the manufacturer) continued after extubation, and if discontinued may be restarted at any time up until ICU discharge. The clinician will have the option of using a loading dose of 1.0 mcg/kg IV over 20 minutes, as recommended by the manufacturer.
  Bedside nursing staff will adjust drug infusion rates as necessary, in consultation with the treating physician, aiming to achieve a Riker Sedation-Agitation Scale 20 score of 4.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Saline placebo — An identical syringe containing only saline with no dexmedetomidine added will be supplied. Initial rate of infusion and subsequent adjustments will be the same as in the active comparator group.
  Arms: Saline placebo

SUMMARY:
The primary aim of the DahLIA trial is to determine, in patients with ICU-associated delirium and agitation who are otherwise pathophysiologically stable (as defined), the number of ventilator-free hours in the incident ICU admission in the 7 days following commencement of trial medication, in patients randomised to receive dexmedetomidine or placebo while receiving all other aspects of standard care.

The null hypothesis assumes no difference in the median number of ventilator-free hours in this ICU admission in the following 7 days, between patients receiving dexmedetomidine and placebo for ICU-associated agitation and delirium.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for the study if, in the opinion of the treating clinician, they continue to require mechanical ventilation only because their degree of agitation requires such a high dose of sedative medication (midazolam or propofol, the only commonly used specific sedatives in our unit) that extubation is not possible, AND in the opinion of their treating intensivist their agitation is so severe as to make lessening their sedation unsafe.

These criteria will be objectively quantified as follows:

* they have required either mechanical restraint and/or anti-delirium or sedative medication in the 4 hours prior to seeking consent AND
* their Confusion Assessment Method for the ICU (CAM-ICU) test is positive for delirium in the 4 hours prior to seeking consent AND
* their Motor Activity Assessment Scale (MAAS) score is 5 or more in the 4 hours prior to seeking consent, confirming psychomotor agitation AND
* their SOFA score is less than or equal to 5 in the 4 hours prior to seeking consent, predicting a mortality or around 5%.

Exclusion Criteria:

* Age less than 18 years old
* Pregnancy or breastfeeding
* Advanced dementia (in the premorbid state requiring professional nursing care)
* Open or closed head injury
* Death is deemed imminent and inevitable
* The patient has previously been enrolled in the DahLIA study
* Patients who could not be extubated, or who would be intubated within the following 48 hours, even if delirium or agitation were corrected. This will include:

  * Patients receiving high dose opioid for analgesia (not sedation) ( > 40 mg/morphine/day)
  * Patients shortly to return to the operating theatre
  * Patients undergoing repeated invasive procedures, in whom it is desirable to maintain deep sedation
  * Patients likely to require ongoing airway protection or control, or ventilatory support (for example, spinal patients with an inadequate vital capacity)
* Known allergy to haloperidol or alpha 2 agonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ventilator-free hours | 7 days following randomisation
  The primary outcome measure for the study will be the number of ventilator-free hours in the incident ICU admission in the 7 days following commencement of trial medication, in patients randomised to receive dexmedetomidine or normal saline placebo while receiving all other aspects of standard care.

SECONDARY OUTCOMES:
Time to ICU discharge | On hospital discharge, or 6 months (whichever is sooner)
Overall ICU length of stay | On hospital discharge, or 6 months (whichever is sooner)
Time to first extubation | On hospital discharge, or 6 months (whichever is sooner)
Time taken to achieve a satisfactory sedation score | 7 days following randomisation
  Time taken to achieve RASS score -2 to +1 and RIKER score 3 or 4
%ICU time spent with a satisfactory sedation score | 7 days following randomisation
  %ICU time spent with RASS -2 to +1 and RIKER 3 or 4
%ICU time spent with a satisfactory delirium score | 7 days following randomisation
  % time spent with a negative CAM-ICU assessment
Time taken to achieve a satisfactory agitation score | 7 days following randomisation
  Time taken to achieve a MAAS score 2-4
%ICU time spent with a satisfactory agitation score | 7 days following randomisation
  %ICU time spent with a MAAS score 2-4
Need for supplementary sedative medication | 7 days following randomisation
  total infusion time, mean hourly dose and total dose of propofol, morphine and midazolam.
Need for mechanical restraint | 7 days following randomisation
  Time to first not requiring restraint and % ICU time spent without mechanical restraint in the 7 days following commencement of trial medication
Need for supplementary antipsychotic medication | 7 days following randomisation
  Number of doses and total mg delivered of haloperidol, olanzapine, quetiapine, or other anti-psychotic medication as prescribed by the treating physician
Need for tracheostomy | On hospital discharge, or 6 months (whichever is sooner)
  Tracheostomy deemed to be necessary by the treating physician, and actually performed.
Acute hospital length of stay | On hospital discharge, or 6 months (whichever is sooner)
  Total duration of admission to the acute hospital, prior to discharge to home or a skilled or unskilled nursing facility.
Discharge destination | On hospital discharge, or 6 months (whichever is sooner)
  Discharge to home, a skilled nursing facility, residential care, a physical rehabilitation facility, or death.
Daily SOFA score | 7 days following randomisation
  Daily SOFA score with recording of the component parts
ICU mortality | On hospital discharge, or 6 months (whichever is sooner)
  ICU mortality
Hospital mortality | On hospital discharge, or 6 months (whichever is sooner)
  Death in the acute care hospital
Duration and rate of vasopressor support | 7 days following randomisation
  total infusion time, and mean hourly dose of noradrenaline and any other inotrope or vasopressor
Need for insertion of a new central venous catheter to facilitate vasopressor / inotropic support | 7 days following randomisation
Requirement for reintubation | On hospital discharge, or 6 months (whichever is sooner)
  Reintubation of the trachea to facilitate airway protection or mechanical ventilation, as indicated in the opinion of the treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Reade, MBBS DPhil, Study Chair — Austin Hospital & University of Melbourne; Rinaldo Bellomo, MD, Principal Investigator — Austin Hospital and University of Melbourne; John Mulder, MBChB, Principal Investigator — Western Hospital, Melbourne; Ben Cheung, MBBS, Principal Investigator — Toowoomba Hospital; Anthony Delaney, MBBS, Principal Investigator — Royal North Shore Hospital; Andrew Davis, MBBS, Principal Investigator — The Alfred; Steve Webb, MBBS, Principal Investigator — Royal Perth Hospital; Michael Bailey, MSc PhD, Principal Investigator — Monash University; Glenn Eastwood, BNurs RN, Principal Investigator — Austin Hospital, Melbourne Australia
Locations (7):
- Australia (7):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Toowoomba Hospital, Toowoomba, Queensland
  - Northern Hospital, Epping, Victoria
  - The Western Hospital, Footscray, Victoria
  - Austin Hospital, Melbourne, Victoria
  - The Alfred Hospital, Prahran, Victoria
  - Royal Perth Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Reade MC, Eastwood GM, Bellomo R, Bailey M, Bersten A, Cheung B, Davies A, Delaney A, Ghosh A, van Haren F, Harley N, Knight D, McGuiness S, Mulder J, O'Donoghue S, Simpson N, Young P; DahLIA Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Effect of Dexmedetomidine Added to Standard Care on Ventilator-Free Time in Patients With Agitated Delirium: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1460-8. doi: 10.1001/jama.2016.2707. PMID 26975647